CLINICAL TRIAL: NCT07046845
Title: Impact of Perelel Trimester-Specific Dietary Supplements vs. Generic Prenatal Supplements on Maternal and Fetal Health Outcomes: A Randomized Controlled Trial
Brief Title: Perelel Prenatal Supplements vs. Generic Prenatal Supplements and Health of Mother and Baby (SUPPORT)
Acronym: SUPPORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Perelel Inc. (Industry)
Responsible Party: Principal Investigator, Hyagriv Simhan, Professor & Executive Vice Chair, OB/GYN/RS, Director, Clinical Innovation in Women's Health, UPMC, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY25020013
Record Dates: First submitted 2025-03-05; First posted 2025-07-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Perelel Prenatal Supplement Group (Active Comparator)
  Interventions: Dietary Supplement: Perelel Prenatal Vitamin
- Generic Prenatal Supplement Group (Active Comparator)
  Interventions: Dietary Supplement: Generic Prenatal Vitamin
- Observational Arm (No Intervention)

INTERVENTIONS:
Dietary Supplement: Perelel Prenatal Vitamin — Daily Perelel prenatal vitamin supplement throughout pregnancy
  Arms: Perelel Prenatal Supplement Group
Dietary Supplement: Generic Prenatal Vitamin — Daily generic prenatal vitamin supplement throughout pregnancy.
  Arms: Generic Prenatal Supplement Group

SUMMARY:
The goal of this clinical trial is to learn if using Perelel-brand prenatal supplements versus a generic prenatal supplement improves the health of the mother and fetus (unborn baby) during pregnancy.

The main question it aims to answer is:

• How does taking Perelel prenatal supplements versus generic prenatal supplements during pregnancy change the nutritional markers in blood samples?

Participants will:

* Take either Perelel or generic prenatal supplements daily throughout pregnancy
* Visit UPMC Magee-Womens Hospital once every trimester of pregnancy for blood draws and answering questionnaires

In an observational part of this study for different participants, researchers will use blood tests and questionnaires only once during the first trimester to compare pregnant women without food insecurity to those with food insecurity.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant with only one baby
2. Identify as having food insecurity
3. Receiving care at a Magee-Womens Hospital associated prenatal practice
4. Less than 12 weeks' of pregnancy

Exclusion Criteria:

1. Currently using prenatal supplement(s)
2. Unborn baby (fetus) identified as having a chromosomal or structural defect
3. Have a condition that prevents absorption of nutrients from food
4. History of medically treated thyroid disorder
5. Ongoing steroid use

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Marker of Maternal Vitamin D Nutritional Status | Through study completion, an average of 30 weeks
  Assay of Serum 25-hydroxyvitamin D3 in Blood Samples
Marker of Maternal Total Folate (RBC) Nutritional Status | Through study completion, an average of 30 weeks
  Assay of Total Folate (RBC) in Blood Samples
Marker of Maternal Total Folate (Serum) Nutritional Status | Through study completion, an average of 30 weeks
  Assay of Total Folate (Serum) in Blood Samples
Marker of Maternal Serum Ferritin Nutritional Status | Through study completion, an average of 30 weeks
  Assay of Serum Ferritin in Blood Samples
Marker of Maternal Serum Vitamin B12 Nutritional Status | Through study completion, an average of 30 weeks
  Assay of Serum Vitamin B12 in Blood Samples
Marker of Maternal Homocysteine Nutritional Status | Through study completion, an average of 30 weeks
  Assay of Homocysteine in Blood Samples
Marker of Maternal Folate Metabolites Nutritional Status | Through study completion, an average of 30 weeks
  Assay of Folate Metabolites in Blood Samples

SECONDARY OUTCOMES:
Symptoms of Nausea and Vomiting in Pregnancy | Through study completion, an average of 30 weeks
  Symptoms of nausea and vomiting will be assessed using the Pregnancy Unique Quantification of Emesis (PUQ-E) questionnaire score. The PUQ-E has a minimum score of 3 and maximum score of 15, with a higher score meaning more severe symptoms.
Symptoms of Depression in Pregnancy | Through study completion, an average of 30 weeks
  Symptoms of depression will be assessed using the Edinburg Postnatal Depression Scale (EPDS) questionnaire. The EPDS has a minimum score of 0 and maximum score of 30, with a higher score meaning more severe symptoms.
Symptoms of Anxiety in Pregnancy | Through study completion, an average of 30 weeks
  Symptoms of anxiety will be assessed using the State-Trait Anxiety Inventory (STAI) questionnaire. The STAI has a minimum score of 20 and maximum score of 80, with a higher score meaning more severe symptoms.
Symptoms of Stress in Pregnancy | Through study completion, an average of 30 weeks
  Symptoms of stress will be assessed using the Perceived Stress Scale-10 (PSS) questionnaire. The PSS has a minimum score of 0 and maximum score of 40, with a higher score meaning more severe symptoms.
Sleep Quality in Pregnancy | Through study completion, an average of 30 weeks
  Sleep quality will be assessed using the Global Sleep Assessment Questionnaire (GSAQ). The GSAQ has a minimum score of 0 and a maximum score of 45, with a higher score meaning worse sleep quality.
General Maternal Wellness in Third Trimester | Through study completion, an average of 30 weeks
  General maternal wellness in the third trimester will be assessed using the 36-item short-form (SF36) survey questionnaire. The SF36 has a minimum score of 0 and maximum score of 3600, with a higher score meaning a more favorable state.
Result of Clinically Reported Lab Tests of Group B Strep Culture in Pregnancy | Through study completion, an average of 30 weeks
  Group B strep culture result will be abstracted from the medical record. The result will be positive, negative, or missing/not obtained. There are no unit of measurements involved.
Muscle Cramping Symptoms - Severity | Through study completion, an average of 30 weeks
  Severity of muscle cramping symptoms will be assessed by asking, "How severe were they?" (Visual Analog Scale [VAS] response). The VAS responses include the options: Not Severe at All, A Little Severe, Somewhat Severe, Moderately Severe, Very Severe, all of which will be scored on a gradient using a slider.
Muscle Cramping Symptoms - Frequency | Through study completion, an average of 30 weeks
  Frequency of muscle cramping symptoms will be assessed by asking, "In the past week how many days did you experience leg cramps?" (0-7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Hyagriv Simhan, MD, Principal Investigator — Magee-Women's Research Institute
Locations (1):
- UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No